CLINICAL TRIAL: NCT03641937
Title: INVSENSOR00011 Clinical Performance Study
Status: Terminated | Type: Interventional
Why Stopped: Protocol procedure did not adequately meet data needs for the study.
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TP-19045A
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Results first posted 2022-01-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Unapproved Device: Yes

ARMS (1):
- INVSENSOR00011 Test group (Experimental): The subjects will be enrolled into the test group and will receive the INVSENSOR00011 investigational sensor.
  Interventions: Device: INVSENSOR00011

INTERVENTIONS:
Device: INVSENSOR00011 — INVSENSOR00011 - investigational sensor that will be placed on the subject's chest and/or back for the duration of the study.

SUMMARY:
This study assesses the investigational sensor's (INVSENSOR00011) performance for detection of subjects' position and posture in bed, along with heart rate and respiratory rate.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old
* Physical status of ASA I or II
* Must be able to read and communicate in English
* Has signed all necessary related documents, e.g. written informed consent, health assessment questionnaire, gender and ethnicity form, confidentiality agreement
* Passed health assessment screening

Exclusion Criteria:

* Subject has any medical condition which in the judgement of the investigator, renders them inappropriate for participation in the study
* Inability to tolerate sitting still or minimal movement for at least 30 minutes
* Nursing female volunteers
* Excluded at the Principal Investigator's discretion
* Refusal to take pregnancy test (for female subjects)
* Positive pregnancy tests for female subjects of child bearing potential.
* Refusal to shave hair off areas where sensors will be applied (male subjects)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2018-07-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Clinical Lab, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | INVSENSOR00011 Test Group
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- INVSENSOR00011 Test Group: The subjects will be enrolled into the test group and will receive the INVSENSOR00011 investigational sensor.
  INVSENSOR00011: investigational sensor that will be placed on the subject's chest and/or back for the duration of the study.
Arm/Group | INVSENSOR00011 Test Group
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 4
  Black or African American | 4
  Hispanic | 1
  Native American | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of INVSENSOR00011's Posture Change Detection
Description: Correctly detected position changes will be marked as True Positive. Missed detections (if any) will be counted. The sensitivity of INVSENSOR00011's posture change detection will be computed as Sensitivity = True Positive/(True Positive+Missed Detection)
Time Frame: Approximately 30 minutes
Population: The protocol required a minimum of 30 subjects to sufficiently evaluate a detection sensitivity for INVSENSOR00011 sensor's posture change detection algorithm. The study was not able to meet this enrollment target and enrolled only 10 subjects, therefore data should be interpreted with caution due to the insufficient sample size. Across 10 enrolled subjects, there were 100 posture and activity related transitions observed (these include right, left, supine, upright and walking events).
Measure: Number; unit: percent aggregate detection sensitivity
Units Other Than Participants: Posture and Activity Related Transitions
Arm/Group | INVSENSOR00011 Test Group
Number analyzed (Participants) | 10
Number analyzed (Posture and Activity Related Transitions) | 100
percent aggregate detection sensitivity | 99

2. Secondary Outcome: Respiratory Rate Detection
Description: When INVSENSOR00011 respiratory rate (RR) readings are available, it will be compared against reference respiratory rate by computing mean and standard deviation of the differences.
Time Frame: Approximately 20 minutes
Population: The protocol required a minimum of 30 subjects to sufficiently evaluate accuracy of the RR parameter. The study was not able to meet this enrollment target, therefore data should be interpreted with caution due to the insufficient sample size. An error analysis was carried out with reference measurements to assess INVSENSOR00011's RR accuracy. Across 10 enrolled subjects, the RR values from the device was compared against the reference RR to compute mean and standard deviation of bias (SDE).
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | INVSENSOR00011 Test Group
Number analyzed (Participants) | 10
breaths per minute | 3.64 (2.94)

ADVERSE EVENTS:
Time Frame: From the time of INVSENSOR00011 application until the sensor(s) is removed, approximately 30 minutes.
Arm/Group | INVSENSOR00011 Test Group
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/37/NCT03641937/Prot_SAP_001.pdf